CLINICAL TRIAL: NCT05919732
Title: Awake Caudal Catheter Infusion Versus General Anesthesia and Single-dose Caudal Injection for Preterm Neonatal Intensive Care Unit (NICU) Patients Undergoing Inguinal Herniorrhaphy.
Brief Title: Awake Caudal Catheter vs General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Gohalem Felema, Anesthesiologist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-03
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Bupivacaine; Dexmedetomidine; Caffeine; Acetaminophen; Propofol; Rocuronium

STUDY DESIGN:
Intervention Model Description: A prospective, blinded, randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: The statistician for the study will generate a randomization table. An unblinded research coordinator will prepare randomization envelopes which will be numbered sequentially and placed in a bin located in the secure medication room in the peri-operative suite.Intra-operatively, neither the anesthesiologist nor the surgeon will be blinded since they are present from the induction of anesthesia until the conclusion of the operation for patient safety. The doctors, nurses and others caring for the infant postoperatively will be blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caudal Infusion (Experimental): Awake continuous caudal infusion.
  Interventions: Drug: Bupivacaine, Dexmedetomidine, Caffeine, Tylenol
- General anesthesia (Active Comparator): General anesthesia and single-dose caudal injection
  Interventions: Drug: Propofol, rocuronium, caffeine, Tylenol, bupivacaine

INTERVENTIONS:
Drug: Bupivacaine, Dexmedetomidine, Caffeine, Tylenol — bupivacaine .3% + 1: 200,000 epinephrine (dose 3mg/kg). Dexmedetomidine 0.5mcg/kg, Caffeine 15mg/kg, rectal Tylenol 30mg/kg
  Arms: Caudal Infusion
Drug: Propofol, rocuronium, caffeine, Tylenol, bupivacaine — propofol 3mg/kg and rocuronium 0.6mg/kg. Caffeine 15mg/kg and rectal Tylenol 30mg/kg.
  single shot caudal with bupivacaine 0.25% + 1:200,000 epinephrine (total dose 2.5mg/kg)
  Arms: General anesthesia

SUMMARY:
It is well established that preterm inguinal hernias discovered in the NICU pose a significant surgical risk due to the associated co-morbid conditions that accompany these patients. Currently, the standard of care in the United States is general anesthesia. There have been studies that have established that elective outpatient repair of inguinal hernias found in the NICU can be safely performed. Patients that are ready for discharge from the NICU will have inguinal hernia repair prior to leaving. Inguinal hernia repair will also be done on those premature infants that are seen in the Nemours surgical clinic. Spinal anesthesia is currently the most common anesthetic procedure used in the surgical treatment of preterm inguinal hernias after general anesthesia. Caudal catheter technique has been proven to safely provide post-operative care of premature infants. The caudal catheter technique involves placement of a small catheter under ultrasound guidance into the caudal epidural canal to allow re-dosing of local anesthetic during the case and has been shown to be safe and effective management in neonates (Somri M, 2007).

DETAILED DESCRIPTION:
This is a prospective, blinded, randomized controlled trial evaluating the effectiveness of awake caudal catheter infusion versus single dose caudal injection and general anesthesia in the surgical management of preterm infant inguinal hernia repair. Spinal anesthesia has been advocated for but highly rejected in the pediatric surgical community due to its high failure rate, which can be up to 28%. Spinal anesthesia is a form of regional anesthesia involving injection of a local anesthetic into the subarachnoid space, via a fine needle, in a single injection. The failure rate has to do with the time constraint of spinal anesthesia, which is approximately 1 hour. It is difficult to perform a bilateral inguinal hernia in that time duration, necessitating a return trip to the operating room for the contralateral side or intubation midway through the surgical case. An alternative to spinal anesthesia that results in an ability to sustain regional anesthetic effect for a longer duration is the caudal catheter infusion. We hypothesize that awake caudal catheter infusion will allow for the following benefits (1) greater than 2 hour anesthetic time via re-dosing which will allow for the completion of the planned surgical procedure (2) exhibit a negligible failure rate (3) minimize post-operative complications that have been associated with general anesthesia in the preterm neonate.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 60 weeks post gestational age born at less than 37 weeks gestational age.
* Patients in the NICU will meet discharge criteria with or without supplemental oxygen prior to surgical scheduling for inguinal hernia repair.

Exclusion Criteria:

* Patient undergoing other invasive procedures (i.e. gastrostomy tube placement, tracheostomy, laser eye treatment)
* Medical condition that would prevent a regional anesthetic from being performed (i.e. bleeding diathesis, vertebral anomalies, and spinal cord injury prior to surgery)
* Contradictions to the prescribed medications in the protocol.

Ages: 23 Weeks to 60 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Bryskin, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- General Anesthesia: General anesthesia and single-dose caudal injection
  Propofol, rocuronium, caffeine, Tylenol, bupivacaine: propofol 3mg/kg and rocuronium 0.6mg/kg. Caffeine 15mg/kg and rectal Tylenol 30mg/kg.
  single shot caudal with bupivacaine 0.25% + 1:200,000 epinephrine (total dose 2.5mg/kg)
Period: Overall Study
Arm/Group | Caudal Infusion | General Anesthesia
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caudal Infusion | General Anesthesia | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational age | 28.4 (3.3) | 30.0 (4.6) | 29.1 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 10 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20
Weight [Mean (Standard Deviation); unit: kg] | 3.6 (1.0) | 3.1 (0.9) | 3.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Return to Baseline Respiratory Function.
Time Frame: Within 24 hours post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
Participants | 11 | 9

2. Primary Outcome: Surgical Completion.
Time Frame: Within 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
Participants | 11 | 9

3. Primary Outcome: Number of Apneic Episodes.
Description: Cessation of breathing by a premature infant that lasts for more than 20 seconds and/or is accompanied by hypoxia or bradycardia.
Time Frame: 24 hours post operative
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
Episodes | 0.1 (0.3) | 0.9 (1.2)

4. Primary Outcome: Number of Bradycardia Events.
Description: heart rate <90.
Time Frame: 24 hours post operative
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
episodes | 0 (0) | 1.0 (2.0)

5. Secondary Outcome: Days to Hospital Discharge From Surgery
Time Frame: up to 10 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
Days | 2 (2) | 1.6 (0.7)

6. Secondary Outcome: Number of Episodes Requiring Post-operative Narcotics Usage.
Time Frame: 24 hours post operative
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
episodes | 0.3 (0.7) | 0 (0)

7. Secondary Outcome: Operative Time.
Time Frame: Intraoperative, up to 100 minutes.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
Minutes | 57 (28) | 53 (33)

8. Secondary Outcome: Participants Requiring Mechanical Ventilation.
Time Frame: After 24 hours post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
Participants | 0 | 0

9. Secondary Outcome: Number of Participants Returning to Full Feeds.
Time Frame: Within 24 hours post operative
Measure: Number; unit: participants
Arm/Group | Caudal Infusion | General Anesthesia
Number analyzed (Participants) | 11 | 9
participants | 11 | 8

ADVERSE EVENTS:
Time Frame: Within 24 hours post-operative
Arm/Group | Caudal Infusion | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT05919732/Prot_SAP_000.pdf